CLINICAL TRIAL: NCT01236300
Title: In Vivo nCLE Study in the Pancreas With Endosonography of Cystic Tumors
Acronym: INSPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Mauna Kea Technologies (Industry); Institut Paoli-Calmettes (Other); Technical University of Munich (Other); Yale University (Other); University of California, Irvine (Other); Mayo Clinic (Other); University of Washington (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MKT-2010-INSPECT; EUSFNA_02 (Other: Mauna Kea Technologies)
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-05

CONDITIONS: Pancreatic Cysts
Keywords: Pancreatic cysts
MeSH Terms: conditions — Pancreatic Cyst | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cellvizio system (Experimental)
  Interventions: Device: Cellvizio needle-based Confocal Laser Endomicroscopy (nCLE) system

INTERVENTIONS:
Device: Cellvizio needle-based Confocal Laser Endomicroscopy (nCLE) system

SUMMARY:
Assess the safety and efficacy of the Cellvizio needle-based Confocal Laser Endomicroscopy (nCLE) system in differentiating benign from malignant and premalignant cysts (e.g. mucinous from non-mucinous cysts)

DETAILED DESCRIPTION:
The primary aim of the study is to define interpretation criteria to differentiate mucinous from non-mucinous cysts and classify more precisely the cysts. Once these criteria have been defined, the diagnostic parameters of nCLE in differentiating the different types of cysts and the reproducibility of these criteria will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an EUSFNA procedure of a pancreatic cyst,
* Patients aged 18 years or older,
* Patients is under surgical consideration for management of the cyst
* Patients have provided written informed consent for the study

Exclusion Criteria:

* Allergy to fluorescein
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irving Waxman, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- nCLE System: Cellvizio needle-based Confocal Laser Endomicroscopy (nCLE) system was performed in patients with Pancreatic cystic lesions (PCL).
Period: Overall Study
Arm/Group | nCLE System
Started | 66
Completed | 66
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | nCLE System
Number analyzed (Participants) | 66
Age, Continuous [Mean (Full Range); unit: years] | 63.1 [27 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity
Description: Using the descriptive criteria of the nCLE images of mucinous vs. non mucinous cysts determined in stage 1, we assessed diagnostic parameters of needle-based confocal laser endomicroscopy of for the detection of pancreatic cystic neoplasia in stage 2.
  For patients who underwent surgery, a gold standard diagnosis was obtained by histopathological diagnosis of the surgical specimen. The local pathologist reviewed the histology slides and selected key areas for high-resolution digital photography. Digital images for all surgical cases were sent to the central pathologist (J.H.) for review.
  In patients who did not undergo surgery, the final diagnosis was established by clinical diagnosis after a review by five investigators. These investigators independently reviewed the patients' clinical factors, cross-sectional image findings, EUS findings and images, and cyst fluid results, and follow-up imaging studies ranging from 10 to 22 months, if available.
Time Frame: October 2011
Population: Among 66 patients, 26 patients who categorized in Stage 1 only used to develop terms for specific findings, 8 patients were excluded due to insufficient information available to make a consensus diagnosis, and 31 patients in Stage 2 were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- nCLE System (Stage 2): Cellvizio needle-based Confocal Laser Endomicroscopy (nCLE) system was performed in patients with Pancreatic cystic lesions (PCL). Stage 2 assessed whether the specific criteria defiend in Stage 1 could identify pancreatic cystic neoplasms (PCN).
Arm/Group | nCLE System (Stage 2)
Number analyzed (Participants) | 31
percentage of participants | 59 [36 to 79]

2. Secondary Outcome: Overall Complication Rate
Description: Assess the safety of nCLE, by recording any possible adverse event or complications occurring during or shortly after the EUSFNA and nCLE procedure
Time Frame: August 2011
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | nCLE System
Number analyzed (Participants) | 66
percentage of participants | 9 [3 to 19]

3. Primary Outcome: Specificity
Description: as for outcome 1
Time Frame: October 2011
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | nCLE System (Stage 2)
Number analyzed (Participants) | 31
percentage of participants | 100 [66 to 100]

4. Primary Outcome: PPV (Positive Predictive Value)
Description: as for outcome 1
Time Frame: October 2011
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | nCLE System (Stage 2)
Number analyzed (Participants) | 31
percentage of participants | 100 [75 to 100]

5. Primary Outcome: NPV (Negative Predictive Value)
Description: as for outcome 1
Time Frame: October 2011
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | nCLE System (Stage 2)
Number analyzed (Participants) | 31
percentage of participants | 50 [26 to 74]

ADVERSE EVENTS:
Time Frame: Patients were contacted one week after procedure by telephone.
Arm/Group | nCLE System
Serious Adverse Events (participants affected / at risk) | 1/66
Other Adverse Events (participants affected / at risk) | 5/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | nCLE System (N=66)
Pancreatitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | nCLE System (N=66)
Pancreatitis (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Intracystic bleeding (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes